CLINICAL TRIAL: NCT00926328
Title: Comparative Efficacy of a Toothpaste That Reduces Plaque and Gingivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-0507-PL-SP-CT-BS
Record Dates: First submitted 2008-09-26; First posted 2009-06-23 (Estimated); Results first posted 2009-06-23 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Gingivitis
Keywords: Gingivitis and Plaque
MeSH Terms: conditions — Gingivitis; Plaque, Amyloid | interventions — Triclosan; Fluorides; hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A -Experimental toothpaste (Active Comparator): triclosan/copolymer/fluoride toothpaste
  Interventions: Drug: Triclosan, fluoride
- B - control toothpaste (Placebo Comparator): sodium fluoride only toothpaste (placebo)
  Interventions: Drug: Fluoride

INTERVENTIONS:
Drug: Triclosan, fluoride — Six Month study, brush twice daily
  Other Names: Colgate Total Advanced Freshening toothpaste
  Arms: A -Experimental toothpaste
Drug: Fluoride — twice daily usage
  Other Names: Crest Cavity Protection toothpaste
  Arms: B - control toothpaste

SUMMARY:
The objective of this study is to evaluate the performance of two toothpastes in controlling established gingivitis and dental plaque in adults.

ELIGIBILITY:
Inclusion Criteria:

* Availability for the six-month duration of the study.
* Good general health.
* Minimum of 20 uncrowned permanent natural teeth (excluding third molars).
* Initial gingivitis index of at least 1.0 as determined by the use of the Loe and Silness Gingival Index.
* Initial plaque index of at least 1.5 as determined by the use of the Quigley and Hein Plaque Index (Turesky Modification).
* Signed Informed Consent Form.

Exclusion Criteria:

* Presence of orthodontic bands.
* Presence of partial removable dentures.
* Tumor(s) of the soft or hard tissues of the oral cavity.
* Advanced periodontal disease (purulent exudate,tooth mobility, and/or extensive loss of
* periodontal attachment or alveolar bone).
* Five or more carious lesions requiring immediate restorative treatment.
* Use of antibiotics any time during the one month prior to entry into the study.
* Participation in any other clinical study or test panel within the one month prior to entry
* into the study.
* Pregnant women or women who are breast feeding.
* Receive a dental prophylaxis in the past two weeks prior to baseline examinations.
* History of allergic to personal care/consumer products or their ingredients.
* Taking any prescription medicines. That might interfere with the study outcome.
* Individuals with an existing medical condition which prohibits them from not eating or drinking for periods up to 4 hours.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Augusto E Boneta, DDS, Principal Investigator — Dental Research Associates
Locations (1):
- Dr. Fernando Autran, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Performed by the Research Department School of Dentistry UPR
Groups:
- Experimental Treatment: triclosan/copolymer/fluoride toothpaste
- Placebo Control: sodium fluoride toothpaste
Period: Overall Study
Arm/Group | Experimental Treatment | Placebo Control
Started | 60 | 60
Completed | 48 | 46
Not Completed | 12 | 14
Not completed — Lost to Follow-up | 12 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Treatment | Placebo Control | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 58 | 116
  >=65 years | 2 | 2 | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 34.72 (8.51) | 35.95 (10.24) | 35.33 (9.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 43 | 88
  Male | 15 | 17 | 32
Region of Enrollment [Number; unit: participants]
  Spain | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Gingivitis Index
Description: Units on a scale 0 to 3 (0 = no inflammation ,
  1 = Mild inflammation-slight change in color and little change in texture 2 = Moderate inflammation-moderate glazing, redness, edema and hypertrophy. Tendency to bleed upon probing.
  3 = Severe inflammation-marked redness and hypertrophy. Tendency to spontaneous bleeding)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Experimental Treatment | Placebo Control
Number analyzed (Participants) | 48 | 46
Units on a scale | 1.00 (0.17) | 1.27 (0.28)
Statistical Analysis 1: Comparison: Experimental Treatment vs Placebo Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

2. Primary Outcome: Plaque Index
Description: Units on a scale 0 to 5 (0 = no plaque, 1 = separate flecks of plaque on the tooth, 2 = a thin continuous band of plaque, 3 = a band of plaque up to one-third of the tooth, 4 = plaque covering up to two thirds of the of the tooth, 5 = plaque covering two-thirds or more of the crown of the tooth)
Time Frame: 6 Months
Population: Per protocol
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Experimental Treatment | Placebo Control
Number analyzed (Participants) | 48 | 46
Units on a scale | 2.22 (0.49) | 2.88 (0.52)
Statistical Analysis 1: Comparison: Experimental Treatment vs Placebo Control; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Experimental Treatment | Placebo Control
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days